CLINICAL TRIAL: NCT00838981
Title: Pharmacotherapy & CM for Opioid and Cocaine Dependence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0705002636; R01DA021264 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Cocaine Dependence
Keywords: Treatment for addiction; Methadone given for opioid dependence; Cocaine; Opiates
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Modafinil; Sugars; Methadone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Modafinil Plus Contingency Magagement (Active Comparator): Modafinil from 200mg up to 400mg plus Contingency Management
  Interventions: Drug: Modafinil; Behavioral: Contingency Management; Drug: Methadone; Behavioral: cognitive behavioral treatment
- Sugar Pill Plus Contingency Management (Placebo Comparator): Placebo: sugar pill
  Interventions: Drug: Sugar Pill; Behavioral: Contingency Management; Drug: Methadone; Behavioral: cognitive behavioral treatment
- Modafinil Plus Voucher Control (Active Comparator)
  Interventions: Drug: Modafinil; Drug: Methadone; Behavioral: cognitive behavioral treatment; Behavioral: Voucher Control
- Sugar Pill Plus Voucher Control (Placebo Comparator)
  Interventions: Drug: Sugar Pill; Drug: Methadone; Behavioral: cognitive behavioral treatment; Behavioral: Voucher Control

INTERVENTIONS:
Drug: Modafinil — Modafinil is started at 200mg on the first day of week 1 (treatment phase) and increased to 400mg by the end of that week. Subjects will continue to receive 400mg/day for the remainder of the study.
  Arms: Modafinil Plus Contingency Magagement; Modafinil Plus Voucher Control
Drug: Sugar Pill — placebo, sugar pill will mirror active drug
  Other Names: Placebo
  Arms: Sugar Pill Plus Contingency Management; Sugar Pill Plus Voucher Control
Behavioral: Contingency Management — Subjects in the CM conditions will earn vouchers for providing cocaine-free urine specimens. Subjects will be informed of the urine test results when available and, for subjects in the CM condition, receive a voucher at that time if the sample is negative. Subjects in the CM condition earn a minimum of $3 for each urine sample they submit that is negative for cocaine. Voucher amounts will escalate by $1 per consecutive clean urine sample submitted up to a maximum of $15 per clean sample.
  Arms: Modafinil Plus Contingency Magagement; Sugar Pill Plus Contingency Management
Drug: Methadone — Subjects will be started on 30 mg of methadone and the dose will be increased as tolerated to reach 60 mg at the end of the first 1-2 weeks of the induction phase. Methadone dosing will bestabilized. During methadone maintenance (weeks 1-11 of treatment phase), subjects continue to receive their maintenance doses of methadone plus modafinil or placebo.
Behavioral: cognitive behavioral treatment — All subjects will receive a manual-guided CBT treatment over the course of their 16-week participation. This manual-guided therapy promotes abstinence through a functional analysis of high-risk situations and coping skills training.
Behavioral: Voucher Control — Subjects in the Yoked-Control condition (YC) will be paired with a CM subject. Subjects in the YC condition will be informed that they will receive vouchers according to an unpredictable schedule, and that they cannot control when they will receive these vouchers or how much they will be worth.
  Arms: Modafinil Plus Voucher Control; Sugar Pill Plus Voucher Control

SUMMARY:
The purpose of this study is to compare the efficacy of the combined treatment modafinil + Contingency Management (CM) to either treatment condition alone or to yoked-controls on cocaine abstinence.

To investigate the role of modafinil-related improvements in memory, impulse control, and attention in mediating cocaine abstinence.

DETAILED DESCRIPTION:
We hypothesize that the treatment group receiving the combination of modafinil + Contingency Management will have significantly lower cocaine use than the other treatment conditions. We also hypothesize that improvements in memory, impulse control, and attention will be a significant contributor to the treatment improvements investigated in Specific Aim #1.

Opioid and cocaine dependence are major problems among veteran and non-veterans and no effective pharmacotherapy exists for cocaine dependence. Methadone has not shown robust effectiveness in reducing cocaine abuse. Thus, new treatments are needed for the individuals who have developed cocaine dependence. This study is designed to test a new pharmacotherapy for cocaine dependence and is a placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female opioid-dependent patients between the ages of 18-65 will be entered into the study. Females must not be pregnant as determined by pregnancy screening, nor breast feeding, and must be using acceptable birth control methods during study participation.
* Current opioid dependence as evidenced by documentation of prior treatment for opioid dependence or signs of withdrawal, self-reported history of opioid dependence for consecutive 12 month period and a positive urine for opiates.
* Subjects must fulfill DSM-IV criteria for opioid and cocaine dependence.
* Subjects must have a history of cocaine use, with a reported street cocaine use of a minimum of 1/2 gram during the preceding 30 days. Additionally, laboratory confirmation of recent cocaine use (positive urine for cocaine) within 2 weeks prior to admission to the study is required.
* Subjects must be treatment-seekers for opioid and cocaine use.

Exclusion criteria:

* Current DSM-IV diagnosis of other drug or alcohol dependence (other than opiates, cocaine, or tobacco)
* History of heart disease, left ventricular hypertrophy, ischemic ECG changes, chest pain, arrhythmia, hypertension.
* History of severe renal, endocrine or hepatic diseases.
* History of psychosis, schizophrenia, or bipolar type I.
* History of seizure disorder.
* Current use of over-the-counter or prescription psychoactive drugs (antidepressant, anxiolytics, antipsychotics, mood stabilizers, psychostimulants).
* Liver function tests (SGOT,SGPT) greater than 3 times normal.
* Current use of modafinil
* Current suicidality
* Pregnancy or breast-feeding;
* Medical contraindication to treatment with study medication (e.g. for modafinil, history of heart disease, ischemic ECG changes, arrhythmia, hypertension).
* Women of child-bearing potential must agree to use other means of birth control and to have a pregnancy test repeated at least once monthly.
* Known allergy to modafinil or methadone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2008-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D.,Ph.D., Principal Investigator — Yale University
Locations (1):
- Department of Veterans Affairs, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult male and female participants were recruited from the Greater New Haven area from May 2008 to March 2014 by word-of-mouth, flyers and from referrals from treatment centers in the local area. The study was conducted in an outpatient clinic of the West Haven VA Hospital.
Pre-assignment Details: After eligibility was determined, participants were randomized to placebo, 200mg up to 400mg of modafinil.The study consisted of three phases that involve: 1) a one or two week "induction" phase, 2) an eleven-week "treatment" phase; and 3) a four week "taper, detoxification or transfer" phase.
Groups:
- Modafinil Plus Contingency Management: Modafinil from 200mg up to 400mg
  Modafinil: Modafinil will be phase in from 200mg to 400mg
- Modafinil Plus Voucher Control: Modafinil from 200mg up to 400mg plus the voucher control
- Placebo Plus Voucher Control: Sugar pill plus voucher control
- Placebo Plus Contingency Management: Sugar pill plus contingency management
Period: Week 1 Days 1-3
Arm/Group | Modafinil Plus Contingency Management | Modafinil Plus Voucher Control | Placebo Plus Voucher Control | Placebo Plus Contingency Management
Started | 26 | 19 | 27 | 19
Completed | 26 | 19 | 27 | 19
Not Completed | 0 | 0 | 0 | 0
Period: Day 4 to Week 11
Arm/Group | Modafinil Plus Contingency Management | Modafinil Plus Voucher Control | Placebo Plus Voucher Control | Placebo Plus Contingency Management
Started | 26 | 19 | 27 | 19
Completed Main Treatment on 400mg | 22 | 13 | 17 | 14
Completed ('Completed' numbers reflect those that completed the post treatment assessments and 'Not Completed' numbers reflect those that did not complete the post treatment assessments.) | 19 | 11 | 16 | 12
Not Completed | 7 | 8 | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Modafinil Plus CM; Modafinil Plus Voucher Control: Modafinil from 200mg up to 400mg
  Modafinil: Modafinil will be phase in from 200mg to 400mg
- Sugar Pill Plus CM; Sugar Pill Plus Voucher Control: Placebo: sugar pill
  Sugar Pill: placebo, sugar pill will mirror active drug
- Total: Total of all reporting groups
Arm/Group | Modafinil Plus CM | Modafinil Plus Voucher Control | Sugar Pill Plus CM | Sugar Pill Plus Voucher Control | Total
Number analyzed (Participants) | 26 | 19 | 19 | 27 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 19 | 19 | 27 | 91
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (10.8) | 41.5 (9.7) | 34.5 (10.2) | 38.2 (11.4) | 38.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 6 | 11 | 33
  Male | 19 | 10 | 13 | 16 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 3 | 4 | 16
  White | 20 | 10 | 14 | 15 | 59
  More than one race | 1 | 5 | 2 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 19 | 19 | 27 | 91

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Positive Urine Tests
Description: thrice weekly urine tests
Time Frame: up to 12 weeks.
Measure: Mean (Standard Deviation); unit: urine tests
Groups:
- Modafinil Plus Voucher Control: Modafinil: Modafinil is started at 200mg on the first day of week 1 (treatment phase) and increased to 400mg by the end of that week. Subjects will continue to receive 400mg/day for the remainder of the study.
  Voucher Control: Subjects in the Yoked-Control condition (YC) will be paired with a CM subject. Subjects in the YC condition will be informed that the
- Sugar Pill Plus Voucher Control: Sugar Pill: placebo, sugar pill will mirror active drug
  Voucher Control: Subjects in the Yoked-Control condition (YC) will be paired with a CM subject. Subjects in the YC condition will be informed that they will receive vouchers according to an unpredictable schedule, and that they cannot control when they will receive these vouchers or how much they will b
Arm/Group | Modafinil Plus Contingency Magagement | Sugar Pill Plus Contingency Management | Modafinil Plus Voucher Control | Sugar Pill Plus Voucher Control
Number analyzed (Participants) | 26 | 19 | 19 | 25
urine tests
  Total Tests | 32 (8.4) | 30.2 (8.6) | 28.1 (11.2) | 31.4 (7.1)
  Cocaine | 17.5 (13.6) | 16.1 (11.4) | 16.9 (10.7) | 15.8 (11.8)
  Heroine | 16.9 (13.4) | 11.9 (10.7) | 12.3 (11.1) | 14 (13.6)
  Any opiate | 17.7 (13.6) | 12.3 (10.6) | 12.5 (11.1) | 14.3 (13.7)

2. Primary Outcome: Average Maximum Days Abstinent
Time Frame: up to 84 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Modafinil Plus Contingency Magagement | Sugar Pill Plus Contingency Management | Modafinil Plus Voucher Control | Sugar Pill Plus Voucher Control
Number analyzed (Participants) | 25 | 19 | 17 | 23
days
  Alcohol | 69 (21) | 58.3 (26.4) | 67.2 (21.9) | 71.8 (19.6)
  Cocaine | 30.9 (28.2) | 32.7 (24.2) | 24.4 (23.3) | 34.7 (32.1)
  Heroine | 40.7 (30.3) | 46.2 (31.1) | 47.6 (33.4) | 48.4 (33.2)
  Any opiate | 31.7 (28) | 37.4 (27.8) | 43.5 (31.3) | 41.4 (32.6)

3. Secondary Outcome: Average Number of Days Using a Substance Within Treatment
Time Frame: up to 90 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Modafinil Plus Contingency Magagement | Sugar Pill Plus Contingency Management | Modafinil Plus Voucher Control | Sugar Pill Plus Voucher Control
Number analyzed (Participants) | 25 | 19 | 17 | 23
days
  Alcohol | 0.32 (.9) | 1.8 (5.2) | 0.06 (0.24) | 0.13 (0.34)
  Cocaine | 19 (19.1) | 15.6 (15.7) | 18.6 (14.3) | 20.3 (20.2)
  Heroin | 13.8 (23.4) | 11.4 (17.6) | 10.2 (15.6) | 11.7 (18.7)
  Opiate | 21.8 (26) | 13.4 (16.8) | 11.9 (16) | 16.4 (23.1)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Modafinil Plus Contingency Magagement | Sugar Pill Plus Contingency Management | Modafinil Plus Voucher Control | Sugar Pill Plus Voucher Control
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/19 | 0/19 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/19 | 0/19 | 0/27
Other Adverse Events (participants affected / at risk) | 11/26 | 8/19 | 5/19 | 6/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Modafinil Plus Contingency Magagement (N=26) | Sugar Pill Plus Contingency Management (N=19) | Modafinil Plus Voucher Control (N=19) | Sugar Pill Plus Voucher Control (N=27)
Disturbed concentration (Psychiatric disorders) | 3 | 2 | 0 | 1
Agitation (Psychiatric disorders) | 4 | 6 | 3 | 1
Tired (General disorders) | 10 | 6 | 5 | 5
Drowsy (General disorders) | 7 | 3 | 2 | 1
Insomnia (General disorders) | 9 | 2 | 4 | 5
Nightmare (General disorders) | 2 | 4 | 0 | 6
Depression (General disorders) | 9 | 4 | 4 | 4
anxiety (Psychiatric disorders) | 8 | 4 | 5 | 2
Numbness (Nervous system disorders) | 5 | 4 | 2 | 2
Headache (General disorders) | 6 | 3 | 4 | 6
Constipation (Gastrointestinal disorders) | 11 | 8 | 3 | 3
Decreased Appetite (Gastrointestinal disorders) | 4 | 3 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No